CLINICAL TRIAL: NCT04183894
Title: Feasibility of Network-Informed Personalized Treatment for Eating Disorders
Brief Title: Personalized Treatment
Acronym: PT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Cheri Levinson, Assistant Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 18.0622
Record Dates: First submitted 2019-11-20; First posted 2019-12-03 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Eating Disorders; Eating Disorder Symptom
Keywords: eating disorder; network analysis; personalized treatment; mobile app
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized Intervention Based on Network (Experimental): Participants will receive personalized interventions based on their personalized network.
  Interventions: Behavioral: Personalized Intervention

INTERVENTIONS:
Behavioral: Personalized Intervention — Participants will receive a personalized intervention based on their personalized network.

SUMMARY:
The Personalized Treatment Study creates an individualized network of symptoms for a participant with a current eating disorder. This network will be used to develop a personalized treatment intervention. This study aims to 1) determine if personalized treatments can be conducted using a network analysis of patient symptoms, and 2) to assess the effectiveness of network-informed personalized treatment for participants with eating disorders.

DETAILED DESCRIPTION:
Cognitive behavioral theory proposes that cognitions, behaviors, affect, and physiological symptoms interact with each other to maintain and exacerbate psychiatric disorders (Beck, 2011). Network theory identifies core symptoms that maintain and promote the spread of ED psychopathology within individuals (Borsboom & Cramer, 2013). Once identified, core "trigger" symptoms can be directly targeted to disrupt the spread or "activation" of ED behaviors, which would help patients achieve full recovery, and ultimately, prevent relapse. One of the main goals of the Personalized Treatment Study is to create an individualized network for a participant with a current eating disorder, which can be used to develop a personalized treatment intervention. Our research questions are: 1) Can a personalized treatment plan be conducted from a network analysis of patient symptoms, and 2) How effective is this personalized treatment based off of a network of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Current eating disorder diagnosis
* at least 18 years of age,
* not actively suicidal,
* not manic,
* not psychotic

Exclusion Criteria:

* No current eating disorder diagnosis,
* younger than 18 years of age,
* active psychosis,
* active mania, or
* actively suicidal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Symptoms | Prior to, during, and after personalized intervention through approximately one year.
  Changes in eating disorder symptoms will be measured at one month, six month, and 1 year follow-up questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

REFERENCES:
- [Background] Beck, J. S. (2011). Cognitive-behavioral therapy. Clinical textbook of addictive disorders, 491, 474-501.
- [Background] Borsboom D, Cramer AO. Network analysis: an integrative approach to the structure of psychopathology. Annu Rev Clin Psychol. 2013;9:91-121. doi: 10.1146/annurev-clinpsy-050212-185608. PMID 23537483
- [Derived] Levinson CA, Williams BM, Christian C, Hunt RA, Keshishian AC, Brosof LC, Vanzhula IA, Davis GG, Brown ML, Bridges-Curry Z, Sandoval-Araujo LE, Ralph-Nearman C. Personalizing eating disorder treatment using idiographic models: An open series trial. J Consult Clin Psychol. 2023 Jan;91(1):14-28. doi: 10.1037/ccp0000785. PMID 36729494
- [Derived] Levinson CA, Hunt RA, Keshishian AC, Brown ML, Vanzhula I, Christian C, Brosof LC, Williams BM. Using individual networks to identify treatment targets for eating disorder treatment: a proof-of-concept study and initial data. J Eat Disord. 2021 Nov 4;9(1):147. doi: 10.1186/s40337-021-00504-7. PMID 34736538